CLINICAL TRIAL: NCT07345546
Title: Association Between Autonomic Nervous System Dysfunction and Choroidal Vascularity Index (CVI) in Patients With Fibromyalgia: A Cross-Sectional Observational Case-Control Study
Brief Title: Association Between Autonomic Dysfunction and Choroidal Vascularity Index in Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Dilara Ekici Zincirci, Medical Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: Fibromiyalgia2
Record Dates: First submitted 2025-12-25; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia; Autonomic Dysfunction
Keywords: fibromiyalgia
MeSH Terms: conditions — Fibromyalgia; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromiyalgia: Adults aged 18-50 years meeting the 2016 ACR criteria for fibromyalgia.
- Healthy Controls: Age- and sex-matched healthy volunteers without fibromyalgia or major systemic/ocular disease.

SUMMARY:
Fibromyalgia is frequently accompanied by autonomic nervous system dysfunction, often characterized by sympathetic predominance. Alterations in ocular microcirculation have been reported in the presence of autonomic dysfunction, including potential reductions in choroidal vascular parameters. This observational study aims to examine the association between autonomic symptom burden and the choroidal vascularity index (CVI), a quantitative marker of choroidal vascular structure derived from optical coherence tomography (OCT), in individuals with fibromyalgia compared with age- and sex-matched healthy controls.

DETAILED DESCRIPTION:
This is a cross-sectional, observational case-control study planned to investigate the relationship between autonomic nervous system dysfunction and choroidal vascularity index (CVI) in patients diagnosed with fibromyalgia according to the 2016 American College of Rheumatology (ACR) criteria. Participants will include adult females and males aged 18-50 years. Demographic and clinical data will be collected, including age, sex, body mass index (BMI), and disease duration.

Autonomic symptom burden will be assessed using the Composite Autonomic Symptom Score 31 (COMPASS-31). Fibromyalgia severity and its impact on daily functioning will be measured using the Revised Fibromyalgia Impact Questionnaire (FIQR). Central sensitization symptoms will be evaluated with the Central Sensitization Inventory (CSI).

All participants will undergo choroidal imaging using optical coherence tomography (OCT; Heidelberg Engineering, Heidelberg, Germany). CVI will be calculated as the ratio of luminal area to total choroidal area. To reduce operator-dependent variability, CVI quantification will be performed using an open-access artificial intelligence-assisted tool designed for choroidal layer analysis (ChoroidAI / choroidometer.com), with standardized image acquisition conditions.

Primary analyses will compare CVI between the fibromyalgia and control groups and evaluate associations between CVI and autonomic symptom burden, fibromyalgia impact, and central sensitization measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years, female or male
* Fibromyalgia group: diagnosis of fibromyalgia according to 2016 ACR criteria
* Ability and willingness to provide written informed consent
* Adequate ocular media clarity suitable for OCT imaging
* Control group: age- and sex-matched healthy volunteers

Exclusion Criteria:

* Ocular exclusions: cataract or other media opacity; glaucoma or optic nerve disease; ocular surface disorders (e.g., dry eye disease); retinal diseases (e.g., diabetic retinopathy, macular disease); ocular surgery or eye/head trauma within the last 3 months; best-corrected visual acuity < 20/20; refractive error > ±3.00 diopters; intraocular pressure > 21 mmHg; use of topical ophthalmic medications
* Systemic/neurologic exclusions: diabetes mellitus; hypertension; hyperlipidemia; thyroid disorders; inflammatory rheumatic/autoimmune diseases; polyneuropathy or neurodegenerative disease; major depressive disorder or anxiety disorder; heavy smoking (>20 cigarettes/day); alcohol or substance dependence; excessive caffeine intake (>2.5 cups/day)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged 18-50 years with fibromyalgia and matched healthy controls recruited from Prof. Dr. Cemil Taşcıoğlu City Hospital in Istanbul, Turkey.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Choroidal Vascularity Index (CVI) | Single assessment at study visit (baseline)
  CVI computed from OCT-derived choroidal images as luminal area / total choroidal area.
Autonomic Symptom Burden (COMPASS-31 total score) | Single assessment at study visit (baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşçıoğlu Şehir Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) underlying the results reported in the primary publication (including COMPASS-31, FIQR, CSI scores and OCT-derived CVI measurements) will be shared upon reasonable request. All shared data will be anonymized/de-identified and will not include any direct identifiers.